CLINICAL TRIAL: NCT01064219
Title: The Effect of Intrauterine Injection of Human Chorionic Gonadotrophins (hCG) on the Endometrial T-regulatory Cells and the Electronmicroscopic Endometrial Characteristics
Brief Title: Intrauterine Human Chorionic Gonadotrophins (hCG) and Endometrial Treg Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Egyptian IVF-ET Center (Other)
Responsible Party: Principal Investigator, Ragaa Mansour, Director, the Egyptian IVF-ET Center, The Egyptian IVF-ET Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: hCG and Treg cells
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2010-12

CONDITIONS: Infertility
Keywords: hCG; Treg cells; implantation; pinopodes; endometrium
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- intrauterine hCG (Experimental): intrauterine injection of 100 hCG followed by endometrial biopsy
  Interventions: Drug: human chorionic gonadotrophin

INTERVENTIONS:
Drug: human chorionic gonadotrophin — intrauterine injection of 100 IU hCG followed by endometrial biopsy .
  Other Names: choriomon

SUMMARY:
Intrauterine injection of hCG around the time of implantation may increase endometrial Treg cells and improve implantation. It has been demonstrated that regulatory T cells expand during pregnancy. hCG was found to be secreted by the embryo immediately after fertilization and has chemoattractant properties to Treg cells.

DETAILED DESCRIPTION:
Aim of the work:

To study the effect of intrauterine injection of human chorionic gonadotrophin on the endometrial T regulatory cells (Treg cells)and the electromicroscopic endometrial characteristics.

Background:

It has been demonstrated that regulatory T cells expand during pregnancy and are present at the feto-maternal interface at very early stages in pregnancy.

Rational:

Intrauterine injection of hCG around the time of implantation may increase endometrial Treg cells and improve implantation.

Methods:

Intrauterine injection of 100 IU hCG will be done followed by endometrial biopsy to check for Treg cells and pinopodes.

ELIGIBILITY:
Inclusion Criteria:

* Male factor infertility
* Ovulatory factor infertility
* Unexplained infertility
* Female age less than 39

Exclusion Criteria:

* Azoospermia
* Tubal factor infertility
* Pelvic endometriosis

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
the presence of Treg cells and pinopodes in the endometrium | 4 weeks

SECONDARY OUTCOMES:
pregnancy rate | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ragaa Mansour, MD,PhD, Principal Investigator — The Egyptian IVF-ET Center
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- See also: Related Info — http://www.cu.edu.eg/english/